CLINICAL TRIAL: NCT04189393
Title: Microbiome Analysis in esoPhageal, PancreatIc and Colorectal CaNcer Patients Undergoing Gastrointestinal Surgery
Acronym: MA-PPING
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-5859
Record Dates: First submitted 2019-11-25; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Gastrointestinal Cancer; Colorectal Cancer; Pancreatic Cancer; Esophageal Cancer; Rectum Neoplasm; Esophageal Neoplasms; Pancreatic Ductal Adenocarcinoma; Colonic Neoplasms; Gastrointestinal Microbiome; Microbiota; Anastomotic Leak
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Four types of samples will be collected for microbiome analysis: saliva, feces, intraoperative mucosal swabs and drain fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MA-PPING is a multicenter prospective observational study that includes patients undergoing surgery for gastrointestinal cancer.

The study aims to map the oral and gut microbiome of patients diagnosed with pancreatic, esophageal or colorectal cancer during their surgical patient journey from the moment of diagnosis until full recovery (three months after surgery).

DETAILED DESCRIPTION:
Rationale: The gut microbiome is the composition of micro-organisms that reside in the gastrointestinal tract. Under normal circumstances, the microbiome is balanced and has a beneficial effect on gut function. However, when the microbiome is stressed i.e. by an operation, patients' health or medication, the composition of the microbiome may change rapidly and the virulence of its micro-organisms can increase fast. Surgery, in particular gastrointestinal surgery, has a disruptive effect on the mucosal gut barrier and may lead to shifts in microbial composition. Also, the underlying surgical disease itself can be characterized by changes in the microbiome. Gastrointestinal cancer is associated with specified alterations of the microbiome, and the presence of certain microbiota is related with carcinogenesis and lymph node involvement.

Anastomotic leakage is a severe complication after gastrointestinal surgery and several animal studies linked microbial shifts to the development of anastomotic leakage. Only a few, small and explorative, human studies investigated the microbiome during surgery and correlated their findings with the development of postoperative complications. However, the majority of these studies only sampled the microbiome intraoperatively. Surgery-related microbial shifts manifest also in the pre- and postoperative phase, therefore, sampling in these phases is crucial. To further understand the changes of the microbiome composition due to gastrointestinal surgery and the relation with postoperative infectious complications, samples should be collected on several time points; before, during, and after surgery. With this study we aim to map the oral and gut microbiome of patients diagnosed with pancreatic, esophageal or colorectal cancer in a time frame ranging from the work-up for an operation until the postoperative phase to assess the changing composition of the microbiome during a surgical patient journey.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven malignancy of the distal esophagus, pancreatic head/corpus, colon or rectum
* Patients undergoing primary elective surgery with construction of an anastomosis of the gastrointestinal tract
* Adult patients above age 18 years
* Written informed consent

Exclusion Criteria:

* History of chronic gastro-intestinal disease e.g. Crohns disease and ulcerative colitis
* Presence of acute gastrointestinal infection
* Chronic use of oral antibiotics (3 months or longer)
* Patients undergoing gastrointestinal surgery for gastrointestinal cancer in acute setting
* Patients undergoing construction of an end/loop colostomy or ileostomy (following primary resection)
* Patients undergoing colon and/ or rectal resection without construction of an anastomosis
* Patients who have insufficient knowledge of the Dutch language
* Patients who are not able to give reliable answers to the questionnaires due to a (mental) disease or (cognitive) condition
* Patients who are not able to collect microbiome samples due to a physical or mental condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are presented/present at the participating hospitals with a proven gastrointestinal malignancy and scheduled for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Compositional changes of the oral and gut microbiome, assessed by alpha-diversity using 16S rRNA (ribosomal ribonucleic acid) sequencing, described in a surgical patient journey from moment of diagnosis until full recovery | 4 months
  Changes of the microbiome composition during the surgical treatment quantified as alpha-diversity by 16S rRNA sequencing. Samples will be collected on 7 moments, starting one month before surgery until three months after surgery.

SECONDARY OUTCOMES:
Compositional changes of the oral and gut microbiome, assessed by beta-diversity using 16S rRNA sequencing, correlated with neo-adjuvant therapy | 1 month
  The effect of neo-adjuvant therapy on microbiome composition quantified as beta-diversity by 16S rRNA sequencing
Compositional changes of the oral and gut microbiome, assessed by beta-diversity using 16S rRNA sequencing, correlated with antibiotic prophylaxis | 1 week
  The effect of (preoperative) antibiotic prophylaxis on microbiome composition quantified as beta-diversity by 16S rRNA sequencing
Compositional changes of the oral and gut microbiome, assessed by beta-diversity using 16S rRNA sequencing, correlated with bowel preparation | 1 week
  The effect of preoperative bowel preparation on microbiome composition quantified as beta-diversity by 16S rRNA sequencing
Compositional changes of the oral and gut microbiome, assessed by beta-diversity using 16S rRNA sequencing, correlated with selective decontamination of the digestive tract (SDD) | 1 week
  The effect of selective decontamination of the digestive tract (SDD) on microbiome composition quantified as beta-diversity by 16S rRNA sequencing
Compositional changes of the oral and gut microbiome, assessed by beta-diversity using 16S rRNA sequencing, correlated to the development of infectious complications (30-day) | 1 month
  The effect of infectious complications (such as anastomotic leakage, sepsis, wound infection, pneumonia and urinary tract infection) on microbiome composition quantified as beta-diversity by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Stefan AW Bouwense, MD PhD, Principal Investigator — Radboud University Medical Center Nijmegen; Martijn WJ Stommel, MD PhD, Principal Investigator — Radboud University Medical Center Nijmegen; Harry van Goor, MD PhD, Principal Investigator — Radboud University Medical Center Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided